CLINICAL TRIAL: NCT00004923
Title: Dose Escalation Trial of Docetaxel Plus Irinotecan in Patients With Advanced Cancer
Brief Title: Docetaxel and Irinotecan in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067606; YALE-HIC-10023; NCI-G00-1700
Record Dates: First submitted 2000-03-07; First posted 2004-04-28 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of docetaxel and irinotecan in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of irinotecan when combined with docetaxel in patients with advanced solid malignancies. II. Determine the dose limiting toxicity of this regimen in these patients. III. Assess any antitumor activity of this regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study of irinotecan. Patients receive docetaxel IV over 1 hour followed immediately by irinotecan IV over 30 minutes on days 1, 8, 15, and 22. Treatment continues every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 1 year, then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 15-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven solid malignancy for which no effective therapy is currently available CNS metastases allowed if CNS disease is stable for at least 4 weeks following completion of surgery and/or radiotherapy

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: At least 3 months Life expectancy: ECOG 0-2 Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.2 mg/dL SGOT and/or SGPT no greater than 1.5 times upper limit of normal (ULN) (no greater than 2.5 times ULN allowed if alkaline phosphatase no greater than ULN) Alkaline phosphatase no greater than 2.5 times ULN (no greater than 4 times ULN allowed if SGOT and/or SGPT no greater than ULN) Renal: Creatinine clearance at least 55 mL/min Other: HIV negative No active infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No concurrent medical condition that would preclude compliance with study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy regimens containing topotecan, irinotecan, or docetaxel At least 4 weeks since other prior chemotherapy (6 weeks since prior nitrosoureas, melphalan, or mitomycin) Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior wide field radiotherapy No prior radiotherapy to greater than 20% of bone marrow Surgery: See Disease Characteristics Recovered from any prior surgery Other: No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 1999-04; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Murren, MD, Study Chair — Yale University
Locations (2):
- United States (2):
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Bennett Cancer Center, Stamford, Connecticut